CLINICAL TRIAL: NCT02150356
Title: Effects of Aleurone-enriched Products on Fasting and Postprandial Glycemic Homeostasis and Lipid Metabolism in High Cardiovascular Risk Subjects
Brief Title: Effects of Aleurone-enriched Products on Cardiovascular Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, rivellese angela, Gabriele Riccardi, Federico II University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ALEURONE Prot 209/2013
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2015-06

CONDITIONS: Glucose and Lipid Metabolism; Incretin Hormones Plasma Levels; Inflammation, Oxidative Stress and Endothelial Function
MeSH Terms: conditions — Inflammation | interventions — aleurone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aleurone (Experimental): Diet based in aleurone-enriched products for a period of 8 weeks.
  Interventions: Other: Aleurone
- Control (Placebo Comparator): Diet based on refined cereal products for a period of 8 weeks.
  Interventions: Other: Control

INTERVENTIONS:
Other: Aleurone — Diet based in aleurone-enriched products for a period of 8 weeks.
  Arms: Aleurone
Other: Control — Diet based on refined cereal products for a period of 8 weeks.
  Arms: Control

SUMMARY:
Very few studies have evaluated the effect of aleurone-enriched grains on cardiovascular risk factors. Price et al.(2010) have shown that 4-week supplementation of aleurone-enriched products (27 g/day of aleurone) increased betaine concentration in plasma whereas reduced homocysteine and LDL-cholesterol levels. Interestingly, aleurone had no effect on total antioxidant status or endothelial function, whereas an improvement of C-reactive protein was observed (Price RK et al, 2012). It is not known whether consumption of more than 27g/day of aleurone-enriched products with higher ferulic acid biodisponibility and longer time of treatment could influence these parameters in individuals with metabolic syndrome. Noteworthy, no studies have investigated the effect of aleurone-enriched products on fasting and postprandial glycemic homeostasis and lipid metabolism. In addition, mechanisms by which aleurone may act in vivo are still unknown.

The aim of this study is to investigate whether 8 weeks supplementation with aleurone-enriched products may influence glucose and lipid metabolism, incretin hormones levels, satiety, inflammation, oxidative stress and endothelial function in overweight/obese subjects with high cardiovascular risk.

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese subjects of both gender
* Age range between 20 and 70 years
* High cardiovascular and metabolic risk profile will be enrolled in the study
* Waist circumference > 102 cm for men, and > 88 cm for women
* At least one of the characteristics of the metabolic syndrome according to the NCEP/ATP III criteria:

  * Fasting triglycerides ≥150 mg/dl
  * High-density lipoprotein cholesterol <40 mg/dl (men)/<50 mg/dl (women)
  * Blood pressure ≥ 130/85 mmHg
  * Fasting glucose ≥100 mg/dl

Exclusion Criteria:

* Age <20 and >70 years
* Fasting triglycerides ≥400 mg/dl
* Fasting cholesterol >270 mg/dl
* Cardiovascular events (myocardial infarction or stroke) during the 6 months prior to the study; established diabetes mellitus or any chronic disease
* Renal and liver failure (creatinine >1.7 mg/dl and ALT/AST >2 times than normal values, respectively)
* Anaemia (Hb <12 g /dl)
* Any chronic disease
* People treated with antihypertensive drugs will have to keep the type and dosage of medication unchanged during the whole study period

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
change in fasting and postprandial insulin levels | 8 weeks after the dietary intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. Clinical Medicine and Surgery, Federico II University, Naples, Italy, Italy

REFERENCES:
- [Derived] Testa R, Salamone D, Rivellese AA, Riccardi G, Vitale M, Giacco R, Costabile G. Improving Oxidative Stress Through a Wheat Aleurone-Rich Diet: Are Short-Chain Fatty Acids Possible Mediators? Nutrients. 2025 Oct 20;17(20):3290. doi: 10.3390/nu17203290. PMID 41156541
- [Derived] Costabile G, Vitale M, Della Pepa G, Cipriano P, Vetrani C, Testa R, Mena P, Bresciani L, Tassotti M, Calani L, Del Rio D, Brighenti F, Napoli R, Rivellese AA, Riccardi G, Giacco R. A wheat aleurone-rich diet improves oxidative stress but does not influence glucose metabolism in overweight/obese individuals: Results from a randomized controlled trial. Nutr Metab Cardiovasc Dis. 2022 Mar;32(3):715-726. doi: 10.1016/j.numecd.2021.12.016. Epub 2021 Dec 29. PMID 35123855